CLINICAL TRIAL: NCT06982456
Title: Effects of Massage, Pressure Release, and Stretching in the Treatment of Cervical Pain: An Algometric Assessment
Brief Title: Manual Therapy Techniques for Cervical Pain: Algometric Evaluation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Angel Martínez Carrasco, Professor Doctor, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M10/2024/519
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Myofascial Pain Syndromes; Massage; Stretching
Keywords: Trigger Points; Pain Measurement; Physical Therapy; Passive Stretching
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial with three parallel groups. Participants will be randomly assigned to Experimental Group 1, Experimental Group 2, or Control Group. The intervention groups will receive manual therapy techniques (superficial massage, deep massage, and pressure release technique), with or without passive stretching, while the control group will undergo only pressure pain threshold evaluations. Algometric measurements will be performed pre-treatment, post-treatment, and during follow-up at one and two weeks after the intervention.
Who Masked: Participant, Outcomes Assessor
Masking Description: Masking: Double (Participant, Outcomes Assessor) Description: Participants will not be informed about the specific nature of the interventions (e.g., which techniques are expected to be more effective). The assessor conducting the post-intervention measurements will be blinded to group allocation. Therapists cannot be blinded due to the hands-on nature of the treatments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group 1 (Experimental): The intervention will consist of superficial massage, deep massage, and the pressure release technique applied to the upper trapezius. Following this, a post-treatment algometric measurement will be taken.
  Experimental Group 1: Will receive only the manual treatment. Follow-up algometric measurements will be performed on the upper trapezius one week and two weeks after the intervention.
  Interventions: Other: Manual Therapy on the Upper Trapezius with or without Passive Stretching
- Experimental Group 2 (Experimental): The intervention will consist of superficial massage, deep massage, and the pressure release technique applied to the upper trapezius. Following this, a post-treatment algometric measurement will be taken.
  Experimental Group 2: Will receive the same manual treatment followed by passive stretching of the upper trapezius. An algometric measurement will be conducted immediately after stretching, as well as follow-up assessments one week and two weeks later.
  Interventions: Other: Manual Therapy on the Upper Trapezius with or without Passive Stretching
- Control Group (Placebo Comparator): Control Group: Will not receive any intervention but will undergo algometric assessments under the same conditions to enable comparisons with the experimental groups.
  Interventions: Other: Manual Therapy on the Upper Trapezius with or without Passive Stretching

INTERVENTIONS:
Other: Manual Therapy on the Upper Trapezius with or without Passive Stretching — The intervention consists of manual therapy techniques applied to the upper fibers of the trapezius muscle, including superficial massage, deep massage, and pressure release technique. In one of the experimental groups, this treatment is followed by passive stretching. The control group receives no intervention. Algometric measurements (pressure pain threshold) are taken before and after the intervention, and at one-week and two-week follow-up points to assess the effectiveness and persistence of the treatment.

SUMMARY:
The main objective of this study is to evaluate the effectiveness of different manual therapy techniques in the treatment of cervical pain related to the upper trapezius muscle.

The intervention will compare the effects of superficial massage, deep massage, and pressure release technique on pain intensity, assessed through algometry.

Additionally, the study aims to determine whether the application of passive stretching following manual treatment leads to a significantly greater reduction in pain compared to groups that do not receive stretching.

Finally, the persistence of treatment effects will be evaluated one and two weeks after the intervention.

DETAILED DESCRIPTION:
Methodological Design:

This study will be conducted with the participation of undergraduate Physiotherapy students who voluntarily wish to take part in the research.

Inclusion Criteria:

Be an undergraduate student in Physiotherapy. Be between 18 and 40 years old. Have experienced cervical pain at least once in their life. Present pain localized in the upper fibers of the trapezius muscle. Voluntarily agree to participate in the study by signing an informed consent form.

Exclusion Criteria:

Suffer from migraines. Have any diagnosed neurological disorders. Have suffered a recent injury or trauma in the cervical region. Have scoliosis or any other relevant spinal pathology. Present any musculoskeletal condition that could interfere with the study outcomes.

The participants will be randomly assigned to three groups: Experimental Group 1, Experimental Group 2, and Control Group.

Procedure:

All participants in the experimental groups will complete a short survey collecting information such as age, sex, and whether they experienced discomfort in the treated area the following day. Baseline pressure pain thresholds will be assessed using algometry (in Kg/cm²) on the upper fibers of the trapezius muscle prior to the intervention.

The intervention will consist of superficial massage, deep massage, and the pressure release technique applied to the upper trapezius. Following this, a post-treatment algometric measurement will be taken.

Experimental Group 1: Will receive only the manual treatment. Follow-up algometric measurements will be performed on the upper trapezius one week and two weeks after the intervention.

Experimental Group 2: Will receive the same manual treatment followed by passive stretching of the upper trapezius. An algometric measurement will be conducted immediately after stretching, as well as follow-up assessments one week and two weeks later.

Control Group: Will not receive any intervention but will undergo algometric assessments under the same conditions to enable comparisons with the experimental groups.

Study Duration:

The total estimated duration of the study is three weeks.

Week 1: Intervention and pre-/post-treatment algometric assessments. Week 2: First follow-up algometric measurement. Week 3: Final algometric measurement.

ELIGIBILITY:
Inclusion Criteria:

* Be an undergraduate student in Physiotherapy.
* Be between 18 and 40 years old.
* Have experienced cervical pain at least once in their life.
* Present pain localized in the upper fibers of the trapezius muscle.
* Voluntarily agree to participate in the study by signing an informed consent form.

Exclusion Criteria:

* Suffer from migraines.
* Have any diagnosed neurological disorders.
* Have suffered a recent injury or trauma in the cervical region.
* Have scoliosis or any other relevant spinal pathology.
* Present any musculoskeletal condition that could interfere with the study outcomes.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-05-19 (Estimated); Primary Completion 2025-06-06 (Estimated); Study Completion 2025-06-13 (Estimated)

PRIMARY OUTCOMES:
PPT - Pressure Pain Threshold | Three weeks
  Pressure Pain Threshold (PPT) measured with an algometer (kg/cm²) on the upper trapezius fibers.
  Measurements will be taken pre-treatment, immediately post-treatment, and at one and two weeks post-intervention.

SECONDARY OUTCOMES:
Brief questionnaire (self-reported). | Time of assessment: The day after the intervention
  Subjective assessment of the discomfort or pain experienced in the treated area the day. post-treatment discomfort report.
Data collection form (demographic questionnaire). | Prior to the intervention (baseline).
  Collection of participant characteristics including age and sex. Do you suffer from neck pain regularly?

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No